CLINICAL TRIAL: NCT05488873
Title: A Randomized, Double-Blind, Placebo-Controlled, Study of Topical Pirenzepine or Placebo for the Prevention of Dose Limiting Chemotherapy Induced Peripheral Neuropathy in Oncology Patients Administered Carboplatin and Paclitaxel
Brief Title: A Study of Topical Pirenzepine or Placebo in Oncology Patients With Chemotherapy Induced Peripheral Neuropathy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: WinSanTor, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WST-PZP-005
Record Dates: First submitted 2022-07-31; First posted 2022-08-05 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Oncology; Peripheral Neuropathy; Chemotherapy; Carboplatin/Paclitaxel
MeSH Terms: conditions — Neoplasms; Peripheral Nervous System Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Experimental): Participants will apply 4 mL QD Placebo topical solution
  Interventions: Drug: Placebo
- WST-057 Active (Experimental): Participants will apply 4 mL QD WST-057 Active topical solution.
  Interventions: Drug: WST-057 Active

INTERVENTIONS:
Drug: WST-057 Active — WST-057 Topical Solution
  Other Names: Active
  Arms: WST-057 Active
Drug: Placebo — Matching Placebo Topical Solution
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled adaptive study of the safety, tolerability, and exploratory efficacy of once-daily topical WST-057 administered for up to 19 weeks (or up to 24 weeks for subjects who experience a chemotherapy dose delay) to subjects who are also receiving 6 cycles (3 weeks apart) of Carboplatin AUC 5-6 and Paclitaxel 175 mg/m2 (with dose adjustment per institutional guidelines permitted).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled adaptive study of the safety, tolerability, and exploratory efficacy of once-daily topical WST-057 administered for up to 19 weeks (or up to 24 weeks for subjects who experience a chemotherapy dose delay) to subjects who are also receiving 6 cycles (3 weeks apart) of Carboplatin AUC 5-6 and Paclitaxel 175 mg/m2 (with dose adjustment per institutional guidelines permitted). A Data Safety Monitoring Committee will review the safety data for all patients upon the completion of the first 10 patients. An interim analysis for safety and futility (primary and secondary endpoints) will be conducted after the first 20 subjects complete the trial. Based on this analysis an additional 20 subjects will be randomized and the power assessed. Depending on the statistical power after 40 subjects complete, a determination will be made as to whether or not to continue the recruitment up to a maximum of 60 subjects' completing the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, ages > 18 years and older.
2. Scheduled to undergo chemotherapy for an advanced or metastatic (stage 3 or 4) solid tumor with carboplatin and paclitaxel for 6 cycles of treatment. Treatment with immunotherapy agents Avastin (bevacizumab) and/or Keytruda (pembrolizumab) is permitted.
3. Ability to sign informed consent and understand the nature of a placebo-controlled trial.
4. ECOG Performance Status (PS) of 0, 1, or 2.
5. Ability to complete patient reported outcome questionnaires by themselves.
6. Life expectancy ≥ 6 months
7. Females should be either not of childbearing potential as a result of surgery or menopause (1 year after onset), or of childbearing potential and must be practicing a highly effective medically acceptable method of contraception (as defined in section 8.4.4.1), including abstinence; hormonal contraceptives (e.g., combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device or intrauterine system; or vasectomy (partner), for at least 1 month before the screening visit and for 1 month after the last dose of study medication. If access or use of a highly effective medically acceptable method of contraception is not achievable, then a combination of barrier methods (e.g., male condom, female condom, cervical cap, diaphragm, contraceptive sponge) is acceptable. Eligible female subjects must also have a negative pregnancy test at the screening and baseline visit.
8. Males must agree to the use an acceptable form of contraception (as defined in section 8.4.4.1) during sexual contact with a pregnant female or a female of childbearing potential while participating in the study (e.g., male condom with diaphragm, male condom with cervical cap, or male condom in association with spermicide).
9. If diabetic, be on stable antidiabetic treatment (> 2 months prior to screening) (oral or injectable antidiabetic therapy and/or lifestyle) that is not anticipated to change during the course of the study, except if medically required.
10. Fluency (oral and written) in the language in which the standardized tests will be administered

Exclusion Criteria:

1. Pre-existing history (with or without current symptoms) in medical history of any type of peripheral neuropathy due to any cause other than prior chemotherapy (diabetes, alcohol, toxins, neurotoxic treatments, hereditary, autoimmune, etc.).
2. Anyone with prior history of severe paclitaxel hypersensitivity (including anaphylaxis) should be excluded from study enrollment. Pre-treatment is per local standard of care guidelines to prevent a paclitaxel hypersensitivity reaction. Absolute Neutrophil Count (ANC) must be at least 1500 cells/mm3 prior to paclitaxel treatment.
3. Currently taking regular pain medications i.e., gabapentin, pregabalin, amitriptyline or duloxetine. (Exception: opioids, given for the short-term treatment i.e., malignant pain is acceptable. Opioids prescribed for neuropathic pain is excluded).
4. Clinically significant active macrovascular disease, including a) myocardial infarction or cerebrovascular event in the prior 6 months, b) angioplasty or stenting of coronary arteries or coronary artery bypass surgery within the past < 12 months (valve replacements are permitted as long as patient has fully recovered from the surgery), c) diagnosis of congestive heart failure of any NY heart class I-IV, d) stable or progressive angina pectoris.
5. Other medical conditions, which in the opinion of the treating physician/allied health professional would make this protocol unreasonably hazardous for the patient.
6. Vitamin E supplementation (2R-α-tocopherol or equivalent) for any reason > 225 IU (approximately 150mg)/day ≤ 30 days prior to randomization.
7. Any of the following: pregnant women, nursing women and men or women of childbearing potential who are unwilling to employ adequate contraception (as defined in section 8.4.4.1).
8. Head or neck cancers.
9. Scheduled to undergo radiation therapy while on study.
10. History of hemorrhagic stroke.
11. Proliferative retinopathy or maculopathy requiring acute treatment.
12. Patients requiring dialysis.
13. Presence of clinically significant peripheral or autonomic neuropathy.
14. Current use local (topical) anesthetics or analgesics including lidocaine, capsaicin, cannabinoid (CBD) oil/products, or compounded topical pharmaceutical agents.
15. Uncontrolled treated/untreated hypertension (systolic blood pressure [BP] ≥ 180 or diastolic BP ≥ 100 at screening).
16. Amputations of lower extremities or presence of foot ulcers.
17. Uncontrolled or untreated hypothyroidism.
18. Active and/or systemic infections (e.g., HIV, hepatitis C, tuberculosis, syphilis), or a history of severe infection during the 30 days prior to screening.
19. Clinically significant gastric emptying abnormality (e.g., severe gastroparesis).
20. Clinically significant urinary retention or an enlarged prostate.
21. Uncontrolled glaucoma.
22. Other clinically significant, active or progressive (over the past 12 months) disease of the cardiovascular, gastrointestinal, pulmonary, renal, dermatologic, neurologic, genitourinary, endocrine, rheumatologic or hematologic systems that, in the opinion of the Investigator, would compromise the subject's participation in the study, might confound the results of the study, or pose additional risk in administering the study drug.
23. New treatment with (< 3 months) vitamins and supplements at the discretion of the PI.
24. Known or suspected history of alcohol or substance abuse (a stable and regular use of medical marijuana for non-neuropathic indications is acceptable).
25. Mental incapacity, unwillingness, or language barrier precluding adequate understanding of or cooperation with the study.
26. Women of childbearing potential must have a negative pregnancy test at screening and baseline and must agree to use adequate contraceptive methods (as defined in section 8.4.4.1) during the study and for 1 month after the last dose of study drug (see inclusion criterion 7).
27. History of allergy or hypersensitivity to anticholinergics or any of the components of the investigational product formulations (pirenzepine, coconut oil, ethanol, dimethyl sulfoxide (DMSO), surfactants, propylene glycol, etc.).
28. History of sensitive skin, as defined by a requirement to use soap and skin products formulated for "sensitive skin," as determined by the Investigator.
29. Currently taking any medicines to treat overactive bladder (anticholinergic agents, such as Gelnique), or antispasmodics.
30. Inability to perform screening or baseline assessments.

    Patients with any condition that could potentially interfere with the conduct of the study or confound efficacy evaluations, including the following as specified in numbers 31 through 38 below:
31. Presence of pain, or any masquerading symptoms presenting as neuropathy including central pain, radiculopathy, painful arthritis, etc., that could interfere with the interpretation of the neuropathy endpoint assessments at the discretion of the PI.
32. Major skin or soft-tissue lesions in the dosing from below the knees to the bottom of both feet, and hands), small lesions (i.e., size of coin) are acceptable. However, topical application of study drug to these areas should be avoided.
33. Exposure to an experimental drug, experimental biologic, or experimental medical device within 3 months before screening.
34. Any open wound(s) and/or sunburn(s) in the dosing area. Subjects who have a wound and/or sunburn at screening that is anticipated to resolve before day -1 can be enrolled.
35. History of a serious skin disease (as determined by the Investigator), such as skin cancer, psoriasis, stasis dermatitis or eczema.
36. Receipt of a tattoo in the dosing area within 12 months of dosing.
37. Known or untreated Lyme disease.
38. Any abnormal or clinically significant lab or test result, collected from the Screening or Baseline visits that in the Investigator's opinion would not make the subject an ideal participant in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2026-04-26 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by hematology and chemistry blood tests. | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Safety will be assessed by observing changes in patients' blood tests when compared to normal lab values/ranges after once daily dosing of WST-057 solution or placebo. The number of participants with treatment-related adverse events as assessed by CTCAEv5.0 will be reported.
Incidence of Treatment-Emergent Adverse Events as assessed by vital signs (blood pressure (diastolic and systolicmmHg), heart rate (beats per minute), respiratory rate (breaths per minute). | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Safety will be assessed by observing changes in vitals signs (from baseline) in patients after daily topical doses of WST-057 solution or placebo. The number of participants with treatment-related adverse events as assessed by CTCAE v5.0 will be reported.
Incidence of Treatment-Emergent Adverse Events as assessed by ECG (measuring P Wave, QRS complex, QT interval) | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Safety will be assessed by observing changes in ECG parameters (from baseline) in patients after daily dosing of WST-057 solution or placebo. The number of participants with treatment-related adverse events as assessed by CTCAE v5.0 will be reported.
Incidence of Treatment-Emergent Adverse Events as assessed by a dermal assessment (Draize score (scale 0.0-4.0) of the dosing area | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Dermal safety will be assessed by observing changes in dermal scores (from baseline) in patients after daily dosing of WST-057 solution or placebo. The number of participants with treatment-related adverse events as assessed by CTCAE v5.0 will be reported.
Incidence of Treatment-Emergent Adverse Events as assessed by physical examination | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Safety will be assessed by observing changes in physical examination findings (from baseline) in patients after daily dosing of WST-057 solution or placebo. The number of participants with treatment-related adverse events as assessed by CTCAE v5.0 will be reported.
Incidence of Treatment-Emergent Adverse Events as assessed by tumor evaluation using RECIST v1.1 | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Safety will be assessed by observing changes in tumor evaluation of radiology using RECIST v 1.1(from baseline) in patients after daily dosing of WST-057 solution or placebo. The number of participants with treatment-related adverse events as assessed by CTCAE v5.0 will be reported.

SECONDARY OUTCOMES:
Visual Analogue Score (VAS) | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Visual Analogue Scale (VAS) is a patient-reported pain rating scale first used by Hayes and Patterson in 1921. Scores are based on self-reported measures of symptoms that are recorded with a single mark placed at one point along a horizontal line 100 mm in length that represents a continuum between the two ends of the scale - "no pain" on the left end of the scale and the "worst imaginable pain" on the right end of the scale.
Neuropathy Total Symptom Score-6 (NTSS-6) | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  The NTSS-6 is a validated (proctored) patient reported outcome tool that assesses intensity and frequency of different pain modalities (aching, burning, prickling & lancinating pain, numbness and allodynia) in patients with neuropathy.
Functional Assessment of Cancer Therapy/Gynecological Oncology Group-Neurotoxicity-13 (FACT/GOG-Ntx-13) | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  The FACT/GOG-Ntx-13 measures the severity and impact of symptoms of neuropathy over the past 7 days. Scores range from 0 to 48, with lower scores indicating more severe neurotoxicity.
Patient-Reported Outcomes Measurement Information System (PROMIS)-physical function (short form) | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  PROMIS Physical Function (PROMIS PF) measures the outcome of patients with musculoskeletal disorders by assessing physical function through a grading scale of activities of daily living. The PROMIS Short Form v2.0 - Physical Function 8c is an 8-item fixed length short form derived from the PROMIS Physical Function item bank. It has a recall period of the past seven days and includes a 5-point scale with three sets of response options. Six capability-framed questions are administered with one set of response options, "Without any difficulty" to "Unable to do," and two disability framed-questions are administered with two sets response options, "Not at all" to "Cannot do" and "No difficulty at all" to "Can't do because of health". Scores on the PROMIS Short Form v2.0 - Physical Function 8c are reported on a T score metric (mean = 50 and SD = 10), with higher scores reflecting better physical functioning.
Thermal Quantitative Sensory Testing (Cold) | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Quantification of thermal thresholds has proven to be useful for the evaluation of small-fiber function. QST for cold perception thresholds on both great toes will be assessed. A reduction in QST thermal threshold has shown to have high diagnostic value in subjects with chemotherapy-associated neuropathies.
Utah Early Neuropathy Score (UENS) | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  UENS is a simple, rapid, and reproducible test targeted to detect early sensory peripheral neuropathy. It includes motor examination, pin sensation, allodynia, hyperesthesia, large-fiber sensation, and deep tendon reflexes. The sensations are reported on 0-, 1-, or 2-point scoring for normal, reduced or absent vibration or reflexes.
Activity and Fear of Falling Measurement (Short FES-I) | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  The Short FES-I is a shortened version of the falls efficacy scale to assess fear of falling. A 7-question method to give a total that will range from 7 (no concern about falling) to 28 (severe concern about falling).
Intraepidermal Nerve Fiber Density | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  IENF density (IENFD) is the gold standard for the diagnostic of small fiber pathology and for measuring small fiber neuropathy.
Hand Dexterity | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  The grooved pegboard test, a timed, validated, sensory-motor, speed test of a patient's ability to place pegs into a slotted board, will be used to quantify the potential changes in hand dexterity in this patient population.
Chemotherapy dose modifications as assessed by percentage of patients requiring dose reductions of chemotherapy. | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Efficacy will be assessed by observing the number of patients requiring dose reductions of chemotherapy due to sensory peripheral neuropathy.
Chemotherapy dose modifications as assessed by the percentage of patients requiring dose delay of chemotherapy. | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Efficacy will be assessed by observing the number of patients requiring dose delays of chemotherapy due to sensory peripheral neuropathy.
Chemotherapy dose modifications as assessed by median duration of delays (days) between chemotherapy treatments. | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Efficacy will be assessed by calculating the median duration of delays (days) between chemotherapy treatments.
Chemotherapy dose modifications as assessed by the percentage of patients requiring replacement or change to initially prescribed chemotherapy (carboplatin/paclitaxel combination). | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Efficacy will be assessed by observing the number of patients requiring replacement or change to initially prescribed chemotherapy.
Chemotherapy dose modifications as assessed by the percentage of patients stopping chemotherapy before treatment is complete. chemotherapy (carboplatin/paclitaxel combination). | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Efficacy will be assessed by observing the number of patients stopping chemotherapy before treatment is complete due to sensory peripheral neuropathy.
Dose limiting neuropathy as assessed by decrease in chemotherapy-induced peripheral sensory neuropathy ≥ Grade 3. | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Efficacy will be assessed by change in chemotherapy-induced peripheral sensory neuropathy ≥ Grade 3 as assessed by the sensory neuropathy item from the Common Terminology Criteria for Adverse Events (CTCAE) v 5.0.
Dose limiting neuropathy as assessed by decrease in percentage of patients with sensory peripheral neuropathy ≥ Grade 3 | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Efficacy will be assessed by a change in the percentage of patients with sensory peripheral neuropathy ≥ Grade 3.
Dose limiting neuropathy as assessed by increase in time to onset of sensory peripheral neuropathy ≥ Grade 3. | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Efficacy will be assessed by a change in the time to onset of sensory peripheral neuropathy ≥ Grade 3; using incidences of the adverse event while the patient was receiving chemotherapy.
Dose limiting neuropathy as assessed by decrease in duration of sensory peripheral neuropathy ≥ Grade 3. | 19 weeks or 24 weeks for subjects on a chemotherapy dose delay
  Efficacy will be assessed by a change in the duration of sensory peripheral neuropathy ≥ Grade 3; using the time from onset of grade 3+ neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hansen, Study Director — WinSanTor, Inc
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No